CLINICAL TRIAL: NCT02793882
Title: Correlation Between SUV on 18F-Fluorocholine PET/CT and Gleason Score in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: 13-047
Record Dates: First submitted 2016-05-23; First posted 2016-06-08 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: 18F-Fluorocholine PET/CT
  Other Names: FCH

SUMMARY:
1.0 Background & Introduction Positron emission tomography / computer tomography (PET/CT) is a nuclear medicine procedure based on the measurement of positron emission from radiolabelled tracers. This technology allows biologic processes to be visualized and measured on whole body images. Common radiotracers in use today in the USA and Europe are radiolabelled choline derivatives such as the analogs 18F-fluoromethylcholine (FMCh) and 18F-fluoroethylcholine (FECh), or more broadly FCH. Both of these fluorinated choline analogs have been extensively studied and display seemingly identical biological, radiopharmaceutical and radiochemical properties. Both have been extensively studied in human prostate cancer, with FMCh having slightly more published data than FECh. Imaging with radiolabelled choline derivatives is used to determine sites of abnormal choline metabolism and can be used to characterize prostate cancer, for which there is extensive data in the literature. PET/CT with radiolabelled choline derivatives is considered standard of care by some experts where available, however at the JGH, anatomic imaging with CT and MRI, and bone scan are the current diagnostic imaging modalities in use for this patient population. Prostate cancer cells have increased choline uptake compared to normal tissues, forming the molecular basis for this technique. The Gleason score, a histopathologic measure of tumor aggressiveness, is one of the most important prognostic factors in the disease. The objective of this study is to evaluate if the degree of uptake measured by maximum standard uptake value (SUVmax) on FCH PET/CT in prostate cancer correlates with Gleason score at initial biopsy.

2.0 Study Objectives The objective of this study is to evaluate if the patient-wide SUVmax on 18F-FCH PET/CT in locoregional and metastatic prostate cancer correlates with histopathologic Gleason score at initial biopsy. It is hypothesized that SUVmax will correlate positively with Gleason score. This is of interest because non-invasive risk stratification may be possible in the future.

3.0 Study Design This will be a single-site JGH-only open label study in which one (1) 18F-FCH PET/CT will be performed on study participants. A PET/CT scan takes about 3 hours.

4.0 Safety & Ethics The radiation dose to patients from fluorinated choline derivatives compares favorably to the major PET tracer in widespread clinical use, 18F-fluorodeoxyglucose (18F-FDG). The safety of fluorinated choline derivatives is not disputed and the investigators expect the number of adverse events in this study to be at (or near) zero. There is no established toxicology for diagnostic doses of fluorinated choline derivatives.

There are no salient ethical considerations identified. The treating physicians are free to order any diagnostic or therapeutic intervention on study patients, and care will not be modified or restricted in any way. Treating physicians are free to incorporate information acquired with this study or discard it if it is not relevant. Care of the patients may be improved with additional information provided by FCH PET/CT, but it is otherwise unchanged. No vulnerable populations will be included in the study.

5.0 Confidentiality All information (medical history, physical examination, and PET/CT results) will be kept strictly confidential and only authorized personnel will have access. The reports of the PET/CT will be contained in a password protected radiology & nuclear medicine RIS database (RadImage) where all other diagnostic imaging reports are securely stored. Clinical PET/CT reports will be stored indefinitely, whereas all other study data will be kept locked by the PI and destroyed after 10 years.

6.0 Population, Sample Size and Recruitment A maximum of 225 competent adult male medically stable prostate cancer patients with available Gleason Scores will be entered into the study. Patients will be recruited by urologists in the clinical setting. Initial contact and consent will be by the department of urology.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18+
* prostate cancer

Exclusion Criteria:

* Claustrophobia

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Competent adult male medically stable prostate cancer patients with available Gleason Scores
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03-25 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Patient-wide SUVmax on 18F-FCH PET/CT in locoregional and metastatic prostate cancer | Immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada